CLINICAL TRIAL: NCT02506153
Title: A Phase III Randomized Trial Comparing Physician/Patient Choice of Either High Dose Interferon or Ipilimumab to MK-3475 (Pembrolizumab) in Patients With High Risk Resected Melanoma
Brief Title: Physician/Patient Choice of Either High-Dose Recombinant Interferon Alfa-2B or Ipilimumab, Versus Pembrolizumab in Treating Patients With Stage III-IV High Risk Melanoma That Has Been Removed by Surgery
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2014-02676; NCI-2014-02676 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1404 (Other: SWOG); S1404 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Results first posted 2024-08-27 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-08

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Cutaneous Melanoma; Metastatic Mucosal Melanoma; Metastatic Non-Cutaneous Melanoma; Non-Cutaneous Melanoma; Recurrent Cutaneous Melanoma; Recurrent Mucosal Melanoma; Recurrent Non-Cutaneous Melanoma
MeSH Terms: conditions — Melanoma | interventions — Specimen Handling; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; pembrolizumab; Introns; Interferon alpha-2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (high-dose recombinant interferon alfa-2B, ipilimumab) (Active Comparator): INDUCTION THERAPY: Patients receive high-dose recombinant interferon alfa-2B intravenously (IV) over 20 minutes on days 1-5. Treatment repeats weekly for 4 weeks in the absence of disease progression or unacceptable toxicity. Or patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 3 weeks for a total of 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive high-dose recombinant interferon alfa-2B subcutaneously (SC) on days 1, 3, and 5. Treatment repeats every 6 weeks for up to 48 weeks in the absence of disease progression or unacceptable toxicity. Or patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 12 weeks for 3 years in the absence of disease progression or unacceptable toxicity.
  Patients undergo CT scan, PET scan, MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Biological: Recombinant Interferon Alfa-2b
- Arm II (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 52 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, PET scan, MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
  Arms: Arm I (high-dose recombinant interferon alfa-2B, ipilimumab)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Arm I (high-dose recombinant interferon alfa-2B, ipilimumab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Arm II (pembrolizumab)
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Recombinant Interferon Alfa-2b — Given IV and SC
  Other Names: Alfatronol; Bioferon; Bioferon (TM); Glucoferon; Heberon Alfa; IFN alpha-2B; Interferon alfa 2b; Interferon Alfa-2B; Interferon Alpha-2b; Intron A; Sch 30500; Urifron; Viraferon
  Arms: Arm I (high-dose recombinant interferon alfa-2B, ipilimumab)

SUMMARY:
This randomized phase III trial studies how well pembrolizumab works compared with the current standard of care, physician/patient choice of either high-dose recombinant interferon alfa-2B or ipilimumab, in treating patients with stage III-IV melanoma that has been removed by surgery but is likely to come back or spread. High-dose recombinant interferon alfa-2B may help shrink or slow the growth of melanoma. Immunotherapy with monoclonal antibodies, such as ipilimumab and pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. It is not yet known whether pembrolizumab is more effective than the current standard of care in treating patients with melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare overall survival (OS) of patients with resected stage III and IV melanoma treated with physician/patient choice of either high dose interferon recombinant interferon alfa-2b (alfa-2b) or ipilimumab versus MK-3475 (pembrolizumab).

II. Among patients who are PD-L1 positive, to compare OS of patients with resected stage III and IV melanoma treated with physician/patient choice of either high dose interferon alfa-2b or ipilimumab versus MK-3475 (pembrolizumab).

III. To compare relapse-free survival (RFS) of patients with resected stage III and IV melanoma treated with physician/patient choice of either high dose interferon alfa-2b or ipilimumab to MK-3475 (pembrolizumab).

SECONDARY OBJECTIVES:

I. To estimate OS and RFS for patients who are PD-L1 negative or PD-L1 indeterminate in this population.

II. To compare OS and RFS of patients between the two arms within PD-L1 positive and negative subgroups and to look at the interaction between PD-L1 (positive versus negative) and treatment arm.

III. To assess the safety and tolerability of the regimens.

ADDITIONAL OBJECTIVES:

I. To bank tissue and whole blood in anticipation of future correlative studies in this patient population.

II. To evaluate PD-L1 expression through immunohistochemistry assay. III. To evaluate the effect of treatment-related side effects that may have an impact on the health-related domains of quality of life (QOL) using the Functional Assessment of Cancer Therapy (FACT)-Biological Response Modifiers (BRM), European Quality of Life Five Dimension Three Level Scale (EQ-5D-3L), and Functional Assessment of Chronic Illness Therapy Diarrhea (FACIT-D) between patients treated with physician/patient choice of either high-dose interferon alfa-2b or ipilimumab and MK-3475 (pembrolizumab).

IV. Pharmacokinetic (PK) and anti-drug antibody (ADA) testing will be performed on all patients receiving MK-3475 (pembrolizumab).

TRANSLATIONAL OBJECTIVES RELATED TO T-CELL RECEPTOR BETA CHAIN SEQUENCING:

I. To evaluate the association between TCR beta variable gene (TRBV) haplotype and grade 3-4 immune-related adverse events (irAEs) among stage III melanoma patients treated with adjuvant ipilimumab or pembrolizumab.

II. To describe the TRBV haplotype distribution among this cohort of patients studied.

TRANSLATIONAL MEDICINAL OBJECTIVE RELATED TO ASSOCIATION OF CIRCULATING TUMOR DNA (ctDNA) WITH RELAPSE-FREE SURVIVAL IN HIGH-RISK, RESECTED MELANOMA PATIENTS.

I. To evaluate associations between pretreatment ctDNA (present versus absent) and relapse within 2 years of randomization in a case-control analysis across treatment arms.

II. To evaluate associations between pretreatment ctDNA (present versus absent) and relapse within 2 years of randomization in a case-control analysis across treatment arms.

III. To evaluate associations between pretreatment ctDNA and relapse within 2 years of randomization in a case-control analysis within each treatment arm (after treatment arm data are unblinded to investigators).

IV. To evaluate associations between "early-on treatment" ctDNA levels and relapse within 2 years of randomization.

V. To describe ctDNA levels at end of therapy and time of relapse.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I:

INDUCTION THERAPY: Patients receive high-dose recombinant interferon alfa-2B intravenously (IV) over 20 minutes on days 1-5. Treatment repeats weekly for 4 weeks in the absence of disease progression or unacceptable toxicity. Or patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 3 weeks for a total of 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive high-dose recombinant interferon alfa-2B subcutaneously (SC) on days 1, 3, and 5. Treatment repeats every 6 weeks for up to 48 weeks in the absence of disease progression or unacceptable toxicity. Or patients receive ipilimumab IV over 90 minutes on day 1. Treatment repeats every 12 weeks for 3 years in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 52 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo computed tomography (CT) scan, positron emission tomography (PET) scan, magnetic resonance imaging (MRI) and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days, 6 and 12 weeks, every 3 months for 2 years, every 6 months for 3 years, and then every 12 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 REGISTRATION:
* Patients must have completely resected melanoma of cutaneous origin or of unknown primary in order to be eligible for this study; patients must be classified as stage IIIA (N2a), IIIB, IIIC, or stage IV melanoma; patients with non-ulcerated T1b N1a disease are not eligible; patients with melanoma of mucosal or other non-cutaneous origin are eligible; patients with melanoma of ocular origin are not eligible; patients with a history of brain metastases are ineligible
* Patients are eligible for this trial either at initial presentation of their melanoma or at the time of the first detected nodal, satellite/in-transit, distant metastases, or recurrent disease in prior lymphadenectomy basin or distant site; nodal, satellite/in-transit metastasis, distant metastases or disease in a prior complete lymphadenectomy basin must have been confirmed histologically by hematoxylin and eosin (H & E) stained slides
* Patients with multiple regional nodal basin involvement are eligible; gross or microscopic extracapsular nodal extension is permitted
* Patients at initial presentation of melanoma must undergo an adequate wide excision of the primary lesion, if present; patients with previously diagnosed melanoma must have had all current disease resected with pathologically negative margins and must have no evidence of disease at the primary site or must undergo re-resection of the primary site; a full lymphadenectomy meeting the criteria outlined is required for all node-positive patients including those with positive sentinel nodes; patients with recurrent disease who have had a prior complete lymphadenectomy fulfill this requirement as long as all recurrent disease has been resected; for all patients, all disease must have been resected with negative pathological margins and no clinical, radiologic, or pathological evidence of any incompletely resected melanoma; patients must be registered within 98 days of the last surgery performed to render the patient free of disease
* Patients must have available and be willing to submit a minimum of five unstained slides from primary, lymph node, or metastatic site to determine PD-L1 expression; the tumor tissue must be adequate for PD-L1 testing (defined as >= 100 tumor cells as confirmed by the treating institution's local pathologist); this must be documented by having a pathologist sign the S1404 Local Pathology Review form prior to step 1 registration; the specimens may come from an archived block but must be submitted within 20 days from cutting the slides
* Patients must be offered the opportunity to participate in specimen banking as outlined
* Patients must be willing to have blood draws for PK/ADA analysis as outlined, should the patient be randomized to the MK-3475 arm
* Patients may have received prior radiation therapy, including after the surgical resection; all adverse events associated with prior surgery and radiation therapy must have resolved to =< grade 1 prior to registration
* Patients must not have received neoadjuvant treatment for their melanoma; patients must not have had prior immunotherapy including, but not limited to ipilimumab, interferon alfa-2b, high dose IL-2, pegylated (PEG)-IFN, anti-PD-1, anti-PD-L1 intra-tumoral, or vaccine therapies; patients must not be planning to receive any of the prohibited therapies during the screening or treatment phases of the study
* Patients must not be planning to receive concomitant other biologic therapy, radiation therapy, hormonal therapy, other chemotherapy, surgery or other therapy after step 2 registration
* All patients must have disease-free status documented by a complete physical examination and imaging studies within 42 days prior to registration; imaging studies must include a total body positron emission tomography (PET)-computed tomography (CT) scan that is of diagnostic quality (with or without brain) or a CT of the chest, abdomen and pelvis; for patients with melanoma arising from the head and neck, dedicated neck imaging (CT with IV contrast or PET-CT through the region) is required; if the patient has had unknown primary with disease in the axilla, neck imaging is required to assure region is clear of cancer; CT imaging should be done with intravenous contrast if there are no contraindications for it; any other clinically-indicated imaging studies if performed (e.g. bone scan) must show no evidence of disease
* All patients must have a CT or magnetic resonance imaging (MRI) of the brain within 90 days prior to registration; the brain CT or MRI should be performed with intravenous contrast (unless contraindicated)
* Absolute neutrophil count (ANC) >= 1,500 microliter (mcL) (within 42 days prior to registration)
* Platelets >= 100,000 mcL (within 42 days prior to registration)
* Hemoglobin >= 10 g/dL (within 42 days prior to registration)
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) (except Gilbert's syndrome, who must have a total bilirubin < 3.0 mg/dL) (within 42 days prior to registration)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2 x IULN (within 42 days prior to registration)
* Alkaline phosphatase =< 2 x IULN (within 42 days prior to registration)
* Serum creatinine =< IULN OR measured or calculated creatinine clearance >= 60 mL/min (within 42 days prior to registration)
* Patients must have lactate dehydrogenase (LDH) performed within 42 days prior to registration
* Patients must have Zubrod performance status =< 1
* Patients must have a baseline electrocardiogram (ECG) performed within 42 days of registration that is normal or considered not clinically significant by the site investigator
* Patients must not have a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Patients must not have an active infection requiring systemic therapy
* Patients must not have active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients must not have received live vaccines within 42 days prior to registration; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, shingles, yellow fever, rabies, bacillus Calmette-Guerin (BCG), and typhoid (oral) vaccine; seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Patients known to be human immunodeficiency virus (HIV) positive are eligible if they meet the following criteria within 30 days prior to registration: stable and adequate cluster of differentiation 4 (CD4) counts (>= 350 mm^3), and serum HIV viral load of < 25,000 IU/ml; patients may be on or off anti-viral therapy so long as they meet the CD4 count criteria
* Patients must not have known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection prior to registration
* Patients must not have a history or current evidence of any condition, therapy or laboratory abnormality that might confound the trial results, interfere with the patient's participation for the full duration of the trial, or indicate that participation in the trial is not in the patient's best interests, in the opinion of the treating investigator
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, lobular carcinoma of the breast in situ, atypical melanocytic hyperplasia or melanoma in situ, adequately treated stage I or II cancer (including multiple primary melanomas) from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years
* Women of childbearing potential must have a negative urine or serum pregnancy test within 28 days prior to registration; women/men of reproductive potential must have agreed to use an effective contraceptive method for the course of the study through 120 days after the last dose of study medication; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy, or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures, he/she is responsible for beginning contraceptive measures; patients must not be pregnant or nursing due to unknown teratogenic side effects
* Patients who are able to complete questionnaires in English, Spanish or French must participate in the quality of life assessments; (those patients who cannot complete the quality of life questionnaires in English, Spanish or French can be registered to S1404 without contributing to the quality of life studies)
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent for this protocol in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* STEP 2 REGISTRATION (RANDOMIZATION CRITERIA):
* Patients must not be registered until receiving confirmation from the Southwest Oncology Group (SWOG) Statistical Center that the patient's tissue specimen was adequate for PD-L1 testing; patients must be registered within 7 working days of receiving the e-mail notification
* Women of childbearing potential must plan to have a urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a negative serum pregnancy test will be required
* No tests or exams are required to be repeated for step 2 registration (randomization); however, patients who are known to have a change in eligibility status after step 1 registration are not eligible for step 2 registration; for example, ANC is not required to be repeated between step 1 and step 2 registration, but the most recent ANC performed before step 2 registration is required to be >= 1,500 mcL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1301 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2026-01-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sapna Patel, Principal Investigator — SWOG Cancer Research Network
Locations (577):
- United States (553):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Virginia G Piper Cancer Care-Del Camino, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - New England Cancer Specialists, Westbrook, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Toledo, Toledo, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Newport Hospital, Newport, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The West Clinic - Wolf River, Germantown, Tennessee
  - The West Clinic - Mid-Town, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (21):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - The Vitalite Health Network - Dr Leon Richard Oncology Centre, Moncton, New Brunswick
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Waterloo Regional Health Network, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Algoma District Cancer Program Sault Area Hospital, Sault Ste. Marie, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Hopital de la Cite-de-la-Sante, Laval, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Ireland (3):
  - Saint Vincent's University Hospital, Dublin, Co Dublin
  - University College Hospital Galway, Galway, Co Galway
  - University Hospital Waterford, Waterford, Co Waterford

REFERENCES:
- [Derived] Unger JM, Darke A, Othus M, Truong TG, Khushalani N, Kendra K, Lewis KD, Faller B, Funchain P, Buchbinder EI, Tarhini AA, Kirkwood JM, Sharon E, Sondak V, Guild SR, Grossmann K, Ribas A, Patel SP. Effectiveness of Adjuvant Pembrolizumab vs High-Dose Interferon or Ipilimumab for Quality-of-Life Outcomes in Patients With Resected Melanoma: A Secondary Analysis of the SWOG S1404 Randomized Clinical Trial. JAMA Oncol. 2023 Feb 1;9(2):251-260. doi: 10.1001/jamaoncol.2022.5486. PMID 36416836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1,301 participants were randomized (SOC arm=654 and Pembrolizumab arm=647). On the SOC arm, 40 participants assigned to HD-IFN didn't receive intervention (36 due to refusal and 4 due to other reasons) and 49 participants assigned to ipilimumab did not receive intervention (41 due to refusal, 2 due to early progression, and 6 due to other reasons). 8 participants assigned to Pembrolizumab didn't receive intervention (4 due to refusal, 2 due to early progression, and 2 due to other reasons).
Groups:
- FDA Approved Regimen (SOC): Participants receive physician/patient choice of either high-dose recombinant interferon alfa-2B (HD-IFN) or Ipilimumab as follows:
  HD-IFN Induction: IV over 20 mins on days 1-5. Tx repeats weekly for 4 weeks in the absence of disease progression or unacceptable toxicity.
  Maintenance: SC on days 1, 3, and 5. Tx repeats every 6 weeks for up to 48 weeks in the absence of disease progression or unacceptable toxicity.
  Ipilimumab Induction: IV over 90 mins on day 1. Tx repeats every 3 weeks for a total of 4 cycles in the absence of disease progression or unacceptable toxicity.
  Maintenance: IV over 90 mins on day 1. Tx repeats every 12 weeks for 3 years in the absence of disease progression or unacceptable toxicity.
- MK-3475 (Pembrolizumab): Participants receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | FDA Approved Regimen (SOC) | MK-3475 (Pembrolizumab)
Started | 654 | 647
Completed | 52 | 366
Not Completed | 602 | 281
Not completed — Adverse Event | 359 | 114
Not completed — Refused unrelated to adverse event | 127 | 18
Not completed — Progression/relapse | 91 | 136
Not completed — Death | 2 | 1
Not completed — Other - not protocol specified | 23 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FDA Approved Regimen (SOC) | MK-3475 (Pembrolizumab) | Total
Number analyzed (Participants) | 654 | 647 | 1301
Age, Continuous [Median (Full Range); unit: years] | 57.0 [18.3 to 86.0] | 55.9 [20.0 to 82.6] | 56.75 [18.3 to 86.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 264 | 523
  Male | 395 | 383 | 778
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic: Yes | 18 | 26 | 44
  Hispanic: No | 617 | 604 | 1221
  Hispanic: Unknown | 19 | 17 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 621 | 622 | 1243
  Race: Black | 5 | 1 | 6
  Race: Asian | 6 | 4 | 10
  Race: Pacific Islander | 1 | 0 | 1
  Race: Native American | 0 | 2 | 2
  Race: Multi-Racial | 4 | 0 | 4
  Race: Unknown | 17 | 18 | 35
Stage [Count of Participants; unit: Participants] — Participants were staged using the following criteria and TNM Definitions for Pathologic Staging:
  Stage IIIA: 1-T4a N2a M0
  Stage IIIB: T1-4a N1-N2b M0 T1b (ulcerated) N1-N2a M0 T2b-4b N1-N2a MO T1-4a.b N2c M0
  Stage IIIC: T1-4b N1-N2b M0 Any T N3 M0
  Stage IV: Any T Any N M1
  Stage IIIA is considered to have the better outcome and Stage IV is considered to have the worse outcome.
  Participants
    IIIA | 69 | 76 | 145
    IIIB | 324 | 311 | 635
    IIIC | 222 | 220 | 442
    IV | 39 | 40 | 79
Performance Status [Count of Participants; unit: Participants] — Zubrod Performance Status scores range from 0 to 1, with higher scores reflecting greater disability.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Participants
    0 | 549 | 541 | 1090
    1 | 105 | 106 | 211
Planned Control Arm Regimen [Count of Participants; unit: Participants]
  High Dose Interferon | 154 | 153 | 307
  Ipilimumab | 465 | 454 | 919
  Enrolled prior to amendment | 35 | 40 | 75
PD-L1 Status [Count of Participants; unit: Participants]
  Positive | 536 | 534 | 1070
  Negative | 93 | 94 | 187
  Indeterminate | 25 | 19 | 44

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Time from date of randomization to date of death due to any cause. Patients known to be alive are censored at date of last contact. The results were presented as 5-year OS estimate.
Time Frame: 5 years after last randomization
Population: The analysis population includes the 1301 participants who were eligible and evaluable (654 in the SOC arm and 647 in the MK-3475 arm).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FDA Approved Regimen (SOC) | MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 654 | 647
percentage of participants | 76 [73 to 80] | 82 [78 to 84]

2. Secondary Outcome: Relapse-free Survival (RFS)
Description: Time from date of randomization to date of first documentation of relapse or death due to any cause. Patients last known to be alive and relapse-free are censored at date of last contact.
Time Frame: 5 years after last randomization
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FDA Approved Regimen (SOC) | MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 654 | 647
percentage of participants | 49 [45 to 53] | 58 [54 to 62]

3. Secondary Outcome: Overall Survival (OS) in Participants Who Are PD-L1 Positive
Description: Time from date of randomization to date of death due to any cause. Patients known to be alive are censored at date of last contact.
Time Frame: 94 months; from study start November 10, 2015 to September 15, 2023
Population: The analysis population includes the 1070 participants who were eligible and evaluable with a PDL-1 positive status (536 in the SOC arm and 534 in the MK-3475 arm).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FDA Approved Regimen (SOC) | MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 536 | 534
percentage of participants | 79 [74 to 82] | 83 [80 to 86]

4. Secondary Outcome: Relapse-free Survival (RFS) in Participants Who Are PD-L1 Positive
Description: as for outcome 2
Time Frame: 5 years after last randomization
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FDA Approved Regimen (SOC) | MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 536 | 534
percentage of participants | 51 [46 to 55] | 60 [56 to 64]

5. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported. CTCAE Version 5.0 was used for all AE reporting.
Time Frame: Randomized patients will be followed until death or 94 months (from study start November 10, 2015 to September 15, 2023), whichever occurs first.
Population: Participants who were eligible and received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Groups:
- FDA Approved Regimen: Participants receive physician/patient choice of either high-dose recombinant interferon alfa-2B (HD-IFN) or Ipilimumab as follows:
  HD-IFN Induction: IV over 20 mins on days 1-5. Tx repeats weekly for 4 weeks in the absence of disease progression or unacceptable toxicity.
  Maintenance: SC on days 1, 3, and 5. Tx repeats every 6 weeks for up to 48 weeks in the absence of disease progression or unacceptable toxicity.
  Ipilimumab Induction: IV over 90 mins on day 1. Tx repeats every 3 weeks for a total of 4 cycles in the absence of disease progression or unacceptable toxicity.
  Maintenance: IV over 90 mins on day 1. Tx repeats every 12 weeks for 3 years in the absence of disease progression or unacceptable toxicity.
Arm/Group | FDA Approved Regimen | MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 565 | 639
Participants
  Abdominal pain | 6 | 2
  Acidosis | 1 | 2
  Acute kidney injury | 2 | 2
  Adrenal insufficiency | 9 | 4
  Alanine aminotransferase increased | 44 | 19
  Alkaline phosphatase increased | 3 | 0
  Anemia | 1 | 1
  Anorexia | 2 | 1
  Anxiety | 2 | 0
  Arthralgia | 4 | 3
  Arthritis | 1 | 0
  Aspartate aminotransferase increased | 33 | 14
  Atelectasis | 1 | 0
  Atrial fibrillation | 1 | 0
  Atrial flutter | 0 | 1
  Autoimmune disorder | 2 | 1
  Back pain | 3 | 0
  Blood and lymphatic system disorders - Other | 1 | 0
  Blood bilirubin increased | 2 | 2
  Blurred vision | 1 | 0
  Bone pain | 1 | 0
  Bronchospasm | 0 | 1
  CPK increased | 5 | 2
  Cardiac disorders - Other, specify | 1 | 0
  Cardiac troponin T increased | 1 | 0
  Colitis | 35 | 13
  Colonic perforation | 1 | 0
  Confusion | 2 | 1
  Cough | 1 | 1
  Creatinine increased | 1 | 0
  Cystitis noninfective | 1 | 0
  Dehydration | 3 | 1
  Depression | 4 | 0
  Diarrhea | 54 | 18
  Dizziness | 1 | 0
  Duodenal ulcer | 1 | 0
  Dyspepsia | 1 | 0
  Dyspnea | 12 | 4
  Encephalitis infection | 2 | 0
  Encephalopathy | 1 | 0
  Endocrine disorders - Other, specify | 4 | 2
  Enterocolitis | 6 | 1
  Enterocolitis infectious | 2 | 1
  Erectile dysfunction | 1 | 0
  Esophagitis | 1 | 0
  Eye disorders - Other, specify | 2 | 1
  Eye pain | 0 | 1
  Facial nerve disorder | 0 | 1
  Fall | 1 | 0
  Fatigue | 30 | 3
  Febrile neutropenia | 2 | 0
  Flu like symptoms | 1 | 1
  Forced expiratory volume decreased | 0 | 1
  GGT increased | 1 | 0
  Gastritis | 2 | 0
  Gastrointestinal disorders - Other, specify | 3 | 0
  General disorders and admin site conditions - Other | 2 | 0
  Generalized muscle weakness | 3 | 0
  Headache | 12 | 3
  Hepatic pain | 0 | 1
  Hepatitis viral | 2 | 0
  Hepatobiliary disorders - Other, specify | 2 | 0
  Hiccups | 0 | 1
  Hyperglycemia | 4 | 7
  Hypersomnia | 1 | 0
  Hypertension | 7 | 2
  Hyperthyroidism | 1 | 1
  Hypertriglyceridemia | 8 | 1
  Hypoalbuminemia | 1 | 0
  Hypokalemia | 3 | 0
  Hyponatremia | 14 | 9
  Hypophosphatemia | 3 | 3
  Hypotension | 2 | 0
  Hypothyroidism | 2 | 0
  Hypoxia | 3 | 2
  Immune system disorders - Other, specify | 1 | 2
  Infections and infestations - Other, specify | 2 | 0
  Infusion related reaction | 1 | 1
  Insomnia | 1 | 0
  Joint effusion | 0 | 1
  Leukemia secondary to oncology chemotherapy | 0 | 1
  Leukocytosis | 1 | 0
  Lipase increased | 5 | 1
  Lower gastrointestinal hemorrhage | 1 | 0
  Lung infection | 1 | 4
  Lymphocyte count decreased | 14 | 3
  Meningitis | 3 | 0
  Metabolism and nutrition disorders - Other, specify | 2 | 1
  Mucositis oral | 0 | 2
  Muscle weakness lower limb | 1 | 0
  Musculoskeletal and connective tiss disorder - Other | 1 | 2
  Myalgia | 5 | 1
  Myocardial infarction | 0 | 1
  Myocarditis | 0 | 1
  Myositis | 1 | 1
  Nausea | 9 | 1
  Nervous system disorders - Other, specify | 4 | 2
  Neuralgia | 2 | 0
  Neutrophil count decreased | 51 | 2
  Pain | 1 | 0
  Pain in extremity | 2 | 0
  Pain of skin | 0 | 1
  Pancreatitis | 3 | 5
  Papulopustular rash | 1 | 1
  Peripheral motor neuropathy | 1 | 0
  Peripheral sensory neuropathy | 1 | 0
  Pharyngitis | 1 | 0
  Pleural effusion | 1 | 0
  Pneumonitis | 5 | 4
  Proctitis | 0 | 1
  Proteinuria | 0 | 1
  Pruritus | 6 | 0
  Rash acneiform | 0 | 2
  Rash maculo-papular | 31 | 9
  Rash pustular | 1 | 0
  Resp, thoracic and mediastinal disorders - Other | 0 | 1
  Respiratory failure | 2 | 0
  Restrictive cardiomyopathy | 1 | 0
  Retinal detachment | 0 | 1
  Retinal tear | 0 | 1
  Seizure | 0 | 1
  Sepsis | 3 | 1
  Serum amylase increased | 1 | 1
  Sinus tachycardia | 1 | 0
  Sinusitis | 0 | 1
  Skin and subcutaneous tissue disorders - Other | 2 | 2
  Skin infection | 1 | 1
  Syncope | 6 | 1
  Tremor | 0 | 1
  Vitreous hemorrhage | 0 | 1
  Vomiting | 9 | 1
  Weight loss | 2 | 0
  Wheezing | 0 | 1
  White blood cell decreased | 19 | 0

ADVERSE EVENTS:
Time Frame: Randomized patients will be followed until death or 94 months (from study start November 10, 2015 to September 15, 2023), whichever occurs first.
Description: CTCAE version 5.0 was used for reporting toxicities and SAEs. There were 565 participants in the standard-of-care group and 639 participants in the pembrolizumab group that were evaluable for AEs.
Groups:
- FDA Approved Regimen: Participants receive physician/patient choice of either high-dose recombinant interferon alfa-2B (HD-IFN) or Ipilimumab as follows:
  HD-IFN Induction: IV over 20 mins on days 1-5. Tx repeats weekly for 4 weeks in the absence of disease progression or unacceptable toxicity.
  Maintenance: SC on days 1, 3, and 5. Tx repeats every 6 weeks for up to 48 weeks in the absence of disease progression or unacceptable toxicity.
  Ipilimumab Induction: IV over 90 mins on day 1. Tx repeats every 3 weeks for a total of 4 cycles in the absence of disease progression or unacceptable toxicity.
  Maintenance: IV over 90 mins on day 1. Tx repeats every 12 weeks for 3 years in the absence of disease progression or unacceptable toxicity.
  89 participants did not receive ant protocol treatment and were not evaluable for adverse events, however they were included in the All-Cause Mortality "at Risk" population.
- MK-3475 (Pembrolizumab): Participants receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
  8 participants did not receive ant protocol treatment and were not evaluable for adverse events, however they were included in the All-Cause Mortality "at Risk" population.
Arm/Group | FDA Approved Regimen | MK-3475 (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 130/654 | 131/647
Serious Adverse Events (participants affected / at risk) | 23/565 | 125/639
Other Adverse Events (participants affected / at risk) | 557/565 | 622/639
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FDA Approved Regimen (N=565) | MK-3475 (Pembrolizumab) (N=639)
Anemia (Blood and lymphatic system disorders) | 0 | 4
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 1 | 2
Myocarditis (Cardiac disorders) | 0 | 3
Sinus bradycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 6
Endocrine disorders-Other (Endocrine disorders) | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Blurred vision (Eye disorders) | 0 | 1
Eye disorders-Other (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 5
Anal hemorrhage (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 10
Diarrhea (Gastrointestinal disorders) | 0 | 12
Enterocolitis (Gastrointestinal disorders) | 2 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 1
Jejunal obstruction (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 5
Proctitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 0 | 2
Flu like symptoms (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 0 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Autoimmune disorder (Immune system disorders) | 1 | 0
Immune system disorders-Other (Immune system disorders) | 0 | 2
Appendicitis (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Encephalitis infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 2
Infections and infestations-Other (Infections and infestations) | 0 | 3
Lung infection (Infections and infestations) | 0 | 5
Prostate infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 8
Soft tissue infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 15
Alkaline phosphatase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 10
Blood bilirubin increased (Investigations) | 0 | 3
CPK increased (Investigations) | 2 | 2
Cardiac troponin I increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 4 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Intracranial hemorrhage (Nervous system disorders) | 0 | 2
Nervous system disorders-Other (Nervous system disorders) | 1 | 2
Seizure (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 2
Pregnancy, puerperium and perinatal conditions-Other (Pregnancy, puerperium and perinatal conditions) | 0 | 3
Confusion (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Renal and urinary disorders-Other (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 9
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Social circumstances-Other (Social circumstances) | 0 | 1
Surgical and medical procedures-Other (Surgical and medical procedures) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Lymphedema (Vascular disorders) | 0 | 1
Peripheral ischemia (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 2
Vascular disorders-Other (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FDA Approved Regimen (N=565) | MK-3475 (Pembrolizumab) (N=639)
Anemia (Blood and lymphatic system disorders) | 129 | 115
Adrenal insufficiency (Endocrine disorders) | 29 | 22
Endocrine disorders-Other (Endocrine disorders) | 52 | 28
Hyperthyroidism (Endocrine disorders) | 19 | 54
Hypothyroidism (Endocrine disorders) | 69 | 143
Blurred vision (Eye disorders) | 36 | 33
Eye disorders-Other (Eye disorders) | 34 | 29
Abdominal pain (Gastrointestinal disorders) | 106 | 87
Colitis (Gastrointestinal disorders) | 54 | 13
Constipation (Gastrointestinal disorders) | 103 | 103
Diarrhea (Gastrointestinal disorders) | 295 | 235
Dry mouth (Gastrointestinal disorders) | 42 | 65
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 34 | 42
Nausea (Gastrointestinal disorders) | 256 | 192
Vomiting (Gastrointestinal disorders) | 110 | 68
Chills (General disorders) | 132 | 55
Edema limbs (General disorders) | 34 | 56
Fatigue (General disorders) | 361 | 429
Fever (General disorders) | 135 | 62
Flu like symptoms (General disorders) | 61 | 43
General disorders and admin site conditions - Other (General disorders) | 33 | 29
Non-cardiac chest pain (General disorders) | 16 | 32
Pain (General disorders) | 51 | 73
Infections and infestations-Other (Infections and infestations) | 34 | 38
Sinusitis (Infections and infestations) | 10 | 39
Upper respiratory infection (Infections and infestations) | 29 | 56
Alanine aminotransferase increased (Investigations) | 222 | 103
Alkaline phosphatase increased (Investigations) | 61 | 49
Aspartate aminotransferase increased (Investigations) | 219 | 128
Blood bilirubin increased (Investigations) | 39 | 44
Creatinine increased (Investigations) | 53 | 72
Investigations-Other (Investigations) | 53 | 65
Lymphocyte count decreased (Investigations) | 59 | 69
Neutrophil count decreased (Investigations) | 112 | 25
Platelet count decreased (Investigations) | 97 | 40
Weight loss (Investigations) | 104 | 38
White blood cell decreased (Investigations) | 96 | 55
Anorexia (Metabolism and nutrition disorders) | 178 | 72
Dehydration (Metabolism and nutrition disorders) | 41 | 21
Hyperglycemia (Metabolism and nutrition disorders) | 85 | 113
Hyperkalemia (Metabolism and nutrition disorders) | 31 | 54
Hypertriglyceridemia (Metabolism and nutrition disorders) | 59 | 75
Hypoalbuminemia (Metabolism and nutrition disorders) | 93 | 58
Hypocalcemia (Metabolism and nutrition disorders) | 51 | 31
Hypoglycemia (Metabolism and nutrition disorders) | 13 | 33
Hypokalemia (Metabolism and nutrition disorders) | 61 | 48
Hyponatremia (Metabolism and nutrition disorders) | 93 | 75
Arthralgia (Musculoskeletal and connective tissue disorders) | 80 | 144
Back pain (Musculoskeletal and connective tissue disorders) | 43 | 54
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 39 | 18
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 21 | 41
Myalgia (Musculoskeletal and connective tissue disorders) | 100 | 98
Pain in extremity (Musculoskeletal and connective tissue disorders) | 48 | 69
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 45
Dizziness (Nervous system disorders) | 103 | 71
Dysgeusia (Nervous system disorders) | 55 | 33
Headache (Nervous system disorders) | 249 | 180
Paresthesia (Nervous system disorders) | 12 | 33
Peripheral sensory neuropathy (Nervous system disorders) | 35 | 37
Anxiety (Psychiatric disorders) | 47 | 58
Depression (Psychiatric disorders) | 47 | 40
Insomnia (Psychiatric disorders) | 84 | 73
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 9 | 33
Cough (Respiratory, thoracic and mediastinal disorders) | 103 | 159
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 87 | 89
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 37 | 90
Sore throat (Respiratory, thoracic and mediastinal disorders) | 33 | 57
Alopecia (Skin and subcutaneous tissue disorders) | 41 | 27
Dry skin (Skin and subcutaneous tissue disorders) | 43 | 54
Pruritus (Skin and subcutaneous tissue disorders) | 176 | 171
Rash acneiform (Skin and subcutaneous tissue disorders) | 37 | 39
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 228 | 209
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 63 | 116
Hypertension (Vascular disorders) | 59 | 112
Hypotension (Vascular disorders) | 33 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT02506153/Prot_SAP_001.pdf